CLINICAL TRIAL: NCT02859428
Title: Disease Natural History and Biomarkers of SPG3A, SPG4 and SPG31
Brief Title: Disease Natural History and Biomarkers of SPG3A, SPG4A, and SPG31
Status: Terminated | Type: Observational
Why Stopped: Investigator left NIH
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160158; 16-N-0158
Record Dates: First submitted 2016-08-06; First posted 2016-08-09 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Hereditary Spastic Paraplegia
Keywords: Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin Fibroblasts

GROUPS / COHORTS (1):
- Patients with hereditary spastic paraplegia (HSP): Patients with hereditary spastic paraplegia types 3A, 4 and 31.

SUMMARY:
Background:

Hereditary spastic paraplegia (HSP) usually progresses slowly. Researchers want to learn more about how its symptoms change over time. They want to look for changes in the blood and cells of people with the most common forms of HSP that might allow them to better understand the disease.

Objectives:

To learn more about common forms of hereditary spastic paraplegia and find out how it progresses over time.

Eligibility:

People age 7 and older with SPG3A, SPG4A, or SPG31

Design:

Participants will have 1 two-hour visit each year for up to 5 years.

At 1 visit, adult participants may have a skin biopsy. An area of skin will be numbed then a tool will remove a small piece of skin.

At all visits, all participants will have a physical exam and blood drawn.

At all visits, participants will do a few tasks like walking quickly and climbing stairs.

Participants can give permission for their skin cells, DNA samples, and data to be used in other studies. The samples and data will have no identifying information.

DETAILED DESCRIPTION:
The Neurogenetics Branch (NGB) within the National Institute of Neurological Disorders and Stroke (NINDS) is conducting a study to evaluate patients with hereditary spastic paraplegia types 3A, 4 and 31. The objective of this study is to understand disease progression in these closely related forms of hereditary spastic paraplegia using validated rating scales such as the Spastic Paraplegia Rating Scale (SPRS), and Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36). We also hope to develop biomarkers that could be used in future treatment trials from human serum and by utilizing transcranial magnetic stimulation (TMS) to determine central motor conduction times and resting motor thresholds.

OBJECTIVES

The primary objective of this protocol is to study the natural history of the most common forms of autosomal dominant hereditary spastic paraplegia. The information obtained from validated rating scales (SPRS and SF-36), TMS, and serum biomarkers, will allow for the development of treatment trials. In some cases, blood or other biologic samples (including skin biopsies) will be obtained for future laboratory studies.

STUDY POPULATION

The number of participants to be enrolled will be set to 300.

DESIGN

This is an observational study of autosomal dominant forms of hereditary spastic paraplegia progression, pathophysiology, and biomarkers.

OUTCOME MEASURES

In this study we will track disease progression using the Spastic Paraplegia Rating Scale (SPRS) and SF-36. Also, we will measure levels of plasma lipids, insulin, leptin, and of certain micro RNAs to investigate their utility as biomarkers. We will utilize TMS (combined with nerve conducting studies) to assess central motor conduction times (CMCT) and resting motor thresholds (RMT).

ELIGIBILITY:
* INCLUSION CRITERIA:
* 7 years or older.
* Proven genetic diagnosis or variant of unknown significance considered by the Principal Investigator (PI) to be likely pathogenic at genomic loci associated with SPG3A, SPG4 and SPG31.
* For the subcomponent involving transcranial magnetic stimulation (TMS) / nerve conduction studies, patients must be greater than or equal to 18 years of age and would be willing to undergo the procedure.

EXCLUSION CRITERIA:

* Adults unable to provide consent or minors without a parent or a guardian.
* Unwillingness to consent for collection of biological samples or their cryopreservation.
* Any bleeding disorder that would prevent or present any danger either during blood extraction or skin biopsy, such hemophilia, or the long-term use of anticoagulants such as Coumadin.
* For the subcomponent of this study involving transcranial magnetic stimulation (TMS), performed with nerve conduction studies:

  * Patients under 18 years of age.
  * Patients withwith implanted devices, such as pacemakers, pumps or stimulators.
  * Patients withor metal in the cranium (excluding dental work) or eye.
  * Patients with known seizure disorder.
  * Patients who are unwilling or unable to participate.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of HSP caused by mutations of known pathological significance or variants of unknown significance at the genomic loci associated with the genes ATL1, SPAST and REEP1.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Spastic Paraplegia Rating Scale (SPRS) | Once a year for five years
  Disease progression as measured by the SPRS and SF-36 scales.
SF-36 | Once a year for five years
  Disease progression as measured by the SPRS and SF-36 scales.

SECONDARY OUTCOMES:
Cortical silent period | Once a year for five years
  Cortical silent period
CMCT, resting motor thresholds, MEP amplitude and MEP latency | Once a year for five years
  CMCT, resting motor thresholds, MEP amplitude and MEP latency
miRNA relative quantity. | Once a year for five years
  miRNA relative quantity.
Fasting Triglycerides, total Cholesterol, HDL and LDL, Leptin, Insulin levels. | Once a year for five years
  Fasting Triglycerides, total Cholesterol, HDL and LDL, Leptin, Insulin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Craig D Blackstone, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Ma YM, Zhao L. Mechanism and Therapeutic Prospect of miRNAs in Neurodegenerative Diseases. Behav Neurol. 2023 Nov 23;2023:8537296. doi: 10.1155/2023/8537296. eCollection 2023. PMID 38058356
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-N-0158.html